CLINICAL TRIAL: NCT04853069
Title: The Impact of Oestrogen Administration on Covid-19 Disease
Brief Title: Oestrogen Treatment for COVID-19 Symptoms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Laboratoires Besins International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-05-099
Record Dates: First submitted 2021-04-06; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: COVID-19; Oestrogen
MeSH Terms: conditions — COVID-19 | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Open label, randomized controlled trial, with patients randomized 1:1 to usual care, or usual care + oestrogen therapy.
  Prior to enrolment, an online CRF will be completed which will confirm that the patient meets the inclusion and exclusion criteria. Randomisation will be undertaken by the statistician in Qatar. Separate randomisation codes will be allocated for patients in Qatar and those in India, and separate randomisation will be performed for males and females. Randomisation will be enclosed in sequentially numbered sealed envelopes (with separate envelopes for males and females). Patients will be allocated to either the treatment or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oestrogen Therapy (Active Comparator): Patients will receive standard care + transdermal 17ß-estradiol gel (3 mg) for ten days.
  Interventions: Drug: Transdermal estradiol gel
- Control Group (No Intervention): Patients will receive only standard care.

INTERVENTIONS:
Drug: Transdermal estradiol gel — Patients will receive standard care +/- (randomsed 1:1) transdermal 17ß-estradiol gel (3 mg; applied to forearm, upper arm and shoulder) for ten days.
  Other Names: oestrogel; estrogel
  Arms: Oestrogen Therapy

SUMMARY:
The aim of this trial is to determine whether oestrogen treatment mitigates disease progression and severity in confirmed COVID19.

DETAILED DESCRIPTION:
It is known that (i) women are relatively protected from the impacts of other respiratory viruses, and that oestrogen may partly mediate this effect (ii) Oestrogen protects rodents from SARS-CoV-1 related mortality (iii) Women are relatively protected from developing or dying from severe COVID-19 and (iv) Postmenopausal women taking oestrogen replacement appear less likely to suffer Covid19-related critical illness. These effects may be mediated through oestrogen-related immunomodulation. In addition, however, 17β estradiol reduces expression of ACE2 (the receptor protein through which SARS-CoV-2 gains cellular entry) in tissues such as the kidney. As such, supplemental oestrogen may represent an effective therapy for Covid19.

We will randomise adult men and postmenopausal women with confirmed Covid19 disease to receive 10 days of transdermal oestrogen (3mg/day). The primary endpoint will be evidence of disease progression, indicated by hospitalisation (mild cases) or need for mechanical ventilation or death within 28 days of randomisation for those hospiatlsied. Secondary outcomes will include hospital mortality, duration of hospital admission, admission to ICU/ HDU facility, ICU/ HDU length of stay, need for renal replacement therapy, receipt and duration of invasive mechanical ventilation, cause-specific mortality and time to being fit for hospital discharge

.

ELIGIBILITY:
Inclusion Criteria:

* Acute Covid-19 disease (PCR-confirmed or clinically diagnosed with high certainty)
* Adult males > 18 years of age OR
* Post-menopausal women (spontaneous amenorrhoea for >12 months in the absence of any other cause)

Exclusion Criteria:

Women:

* taking oestrogen supplements or oestrogen receptor antagonists
* with abnormal genital bleeding
* with a history of breast cancer
* with a history of endometrial or ovarian cancer
* with untreated endometrial hyperplasia

Men:

• taking hormone therapies (e.g. for prostate cancer)

Any subject:

* failure to obtain consent
* taking lamotrigine
* with a thromboembolic disorder (e.g. Protein C or Protein S deficiency, antithrombin III deficiency)
* with pre-existing liver or renal disease
* with known allergy to exogenous oestrogens
* with a history of porphyria
* with a history of thromboembolic event including deep vein thrombosis, thromboembolic stroke or pulmonary emboli
* taking part in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-05-17 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Evidence of disease progression for mild cases | 28 days
  Proportion hospitalised within 28 days
Evidence of disease progression in hospitalised patients (moderate and severe cases) | 28 days
  Proportion requiring mechanical ventilation or dying within 28 days

SECONDARY OUTCOMES:
Hospital mortality | 28 days
  Rate of mortality
Duration of hospital admission | 28 days
  Length of stay at hospital
Admission to ICU/ HDU facility | 28 days
  Length of stay at ICU/HDU facility
Need for renal replacement therapy | 28 days
  Proportion requiring renal replacement therapy
Ventilation | 28 days
  Proportion requiring mechanical ventilation within 28 days
Time to being fit for hospital discharge | 28 days
  Time of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar